CLINICAL TRIAL: NCT00519792
Title: Phase Ib Dose Escalation Study of the Safety, Tolerability, Pharmacokinetics and Antiviral Activity of Omega DUROS® and Ribavirin in Subjects With Chronic Hepatitis C Previously Treated With Pegylated Interferon and Ribavirin
Brief Title: Phase 1b Study of Omega DUROS® in Patients With Chronic Hepatitis C Who Relapsed After Prior Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Intarcia Therapeutics (Industry)
Responsible Party: Intarcia Therapeutics, Inc, Intarcia Therapeutics, Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITCA 638-CLP-08
Record Dates: First submitted 2007-08-21; First posted 2007-08-23 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Chronic Hepatitis C
Keywords: Relapse; HCV; Hepatitis C; Interferon; Ribavirin
MeSH Terms: conditions — Hepatitis C, Chronic; Recurrence; Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Omega DUROS: Dose 25
  Interventions: Drug: Omega DUROS device
- 2 (Experimental): Omega DUROS: Dose 50
  Interventions: Drug: Omega DUROS device

INTERVENTIONS:
Drug: Omega DUROS device — Omega DUROS device 25mcg inserted SC for 48 weeks Omega DUROS device 50mcg inserted SC for 48 weeks

SUMMARY:
Omega DUROS® is an implantable drug delivery system designed to deliver omega interferon subcutaneously at a constant rate for 90 days.

This study is being performed to evaluate the safety and antiviral effects of omega interferon delivered by the Omega DUROS® device in combination with ribavirin in subjects with chronic Hepatitis C genotype 1.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Hepatitis C with HCV genotype 1 infection
* Relapse following an end of treatment response after treatment with a pegylated interferon and ribavirin.

Exclusion Criteria:

* Presence or history of non-HCV chronic liver disease
* Treatment with any interferon subsequent to the relapse with pegylated interferon-alpha and ribavirin
* Decompensated liver disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Safety | Week 52

CONTACTS AND LOCATIONS:
Locations (8):
- United States (7):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - St. Louis University, St Louis, Missouri
  - Weill Cornell Medical College, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Liver Institute at Methodist Dallas, Dallas, Texas
  - Alamo Medical Research, San Antonio, Texas
- Fundacion de Investigacion de Diego, San Juan, Puerto Rico